CLINICAL TRIAL: NCT01902862
Title: Pilot Study With Bortezomib in Combination With Rituximab Standard Therapy in Patients With Relapsed or Refractory Follicular Lymphoma and at Least 2 Previous Therapies
Brief Title: An Efficacy and Tolerability Study of Bortezomib in Combination With Rituximab Standard Therapy in Participants With Relapsed or Refractory Follicular Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruitment too slow
Sponsor: Janssen-Cilag G.m.b.H (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR010342; 26866138LYM2021; 2005-003949-14
Record Dates: First submitted 2013-06-07; First posted 2013-07-18 (Estimated); Last update posted 2014-04-01 (Estimated); Status verified 2014-03

CONDITIONS: Lymphoma, Follicular
Keywords: Lymphoma, follicular; Bortezomib; Rituximab
MeSH Terms: conditions — Lymphoma, Follicular | interventions — Bortezomib; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bortezomib plus rituximab (Experimental): Bortezomib will be administered as intravenous infusion as 1.6 milligram per meter square (mg per m^2) on Days 1, 8, 15 and 22 of cycle 1 and Days 36, 43, 50, 57 of cycle 2 and (if applicable) on Days 71, 78, 85, and 92 of Cycle 3. Rituximab will be administered as intravenous infusion as 375 mg per m^2 on Days 36, 43, 50, 57 of cycle 2 and (if applicable) on Days 71, 78, 85, and 92 of Cycle 3.
  Interventions: Drug: Bortezomib; Drug: Rituximab

INTERVENTIONS:
Drug: Bortezomib — Bortezomib will be administered as intravenous infusion as 1.6 milligram per meter square (mg per m^2) on Days 1, 8, 15 and 22 of cycle 1 and Days 36, 43, 50, 57 of cycle 2 and (if applicable) on Days 71, 78, 85, and 92 of Cycle 3.
  Other Names: VELCADE
Drug: Rituximab — Rituximab will be administered as intravenous infusion as 375 mg pert m^2 on Days 36, 43, 50, 57 of cycle 2 and (if applicable) on Days 71, 78, 85, and 92 of Cycle 3.

SUMMARY:
The purpose of this study is to evaluate the efficacy (effectiveness) and tolerability (how well a participant can stand a particular medicine or treatment; ability to be used) of bortezomib in combination with rituximab standard therapy (medicine or medical care given to a participant for a disease or condition) in participants with relapsed or refractory (not responding to treatment) follicular lymphoma (a cancer of the lymph nodes [or tissues] in follicle).

DETAILED DESCRIPTION:
This is a prospective (study following participants forward in time), open-label (all people know the identity of the intervention), multi-center (conducted in more than 1 center), non-randomized (study drug not assigned by chance), single-arm study in participants with relapsed or refractory cluster of differentiation 20 plus (CD-20+) follicular Grade 1 or 2 lymphoma Stage III or IV with at least 2 previous lines of therapy. The study will include 2 phases: a Screening phase and a Treatment phase. The Screening phase will be conducted 2 weeks before the Treatment phase. The Treatment phase will include 3 cycles. The duration of each cycle will be 5 weeks (35 days). After the second cycle, a response will be evaluated. In case of complete response (CR), participants will be followed-up for a period of 1 year. In case of progressive disease (PD), the participant will be excluded from the study, and in case of stable disease (SD) or partial response (PR), an additional cycle of 5 weeks will be applied and a follow-up of 1 year will be performed. In each cycle, participants will receive 1.6 milligram per meter square (mg per m^2) of bortezomib as intravenous (through a vein in the body) infusion (a fluid or a medicine delivered into a vein by way of a needle) on Days 1, 8, 15, 22 of Cycle 1, Days 36, 43, 50 and 57 of Cycle 2 and on Days 71, 78, 85 and 92 of Cycle 3 (if applicable). Cycle 3 will be applicable only in case of SD or PR according to remission criteria after Cycle 2. In Cycles 2 and (if applicable) 3, injection of bortezomib followed by administration of rituximab (in a dose of 375 mg per m^2) will be given as intravenous infusion. If neuropathy (a disturbance in the function of the brain or spinal cord that may affect the nerves and muscles of the body) grade of more than or equal to 2 will occur then a dose of bortezomib will be reduced from 1.6 mg per m^2 to 1.3 mg per m^2 and then to 1.0 mg per m^2. Participants will be analyzed for time to disease progression or relapse, disease free survival, overall survival and remission (when a medical problem gets better or goes away at least for a while) status. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants with histologically confirmed relapsed or refractory follicular Stage III or IV, Grade 1 and 2, cluster of differentiation 20 plus (CD20+) lymphoma (WHO - World Health Organization) that requires therapy
* Participants in whom treatment with rituximab is planned after greater than or equal to 2 cytostatic (inhibition of cell growth) previous therapies
* Women must be either postmenopausal or sterilized; negative pregnancy test at Screening
* Participants with total bilirubin below 1.5-fold upper limit of normal (ULN) and creatinine below 2-fold ULN
* Participants with Karnofsky Status greater than or equal to 60 percent

Exclusion Criteria:

* Participants with previous treatment with bortezomib within 6 months before enrollment or previous treatment with a combination of rituximab and bortezomib
* Participants with previous known allergic reaction to bortezomib, boron or mannitol
* Participants with life-expectancy of less than 3 months
* Participants with malignant neoplasm (cancerous - new growth that is not normal; tumor) (except basalioma) within previous 5 years
* Participants with peripheral (not central) neuropathy (a disturbance in the function of the brain or spinal cord that may affect the nerves and muscles of the body) common terminology criteria for adverse events (CTCAE) grade greater than or equal to 2

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2006-02; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Time to Progression or Relapse | Start of treatment (Day 1 of Cycle 1) up to Month 15
  Time to disease progression is defined as the time from start of treatment to the time of first documentation of disease progression.

SECONDARY OUTCOMES:
Maximum Tolerated Dose (MTD) of Bortezomib in Combination With Rituximab | Start of treatment (Day 1 of Cycle 1) up to Month 15
  MTD is defined as the dose level combination below the dose level that produces a dose-limiting toxicity. If MTD is not reached, the recommended MTD is the maximum dose that the participants received. Tolerability of bortezomib in combination with rituximab standard therapy will be monitored.
Number of Participants With Remission Status | Start of treatment (Day 1 of Cycle 1) up to Month 15
  Participants with complete response (CR), partial response (PR) and stable disease (SD) separately for each category as well as participants with CR or PR (cumulative, i.e., either CR or PR) or participants with CR, PR or SD (cumulative, i.e., either CR or PR or SD) as best remission status will be reported.
Disease-Free Survival | Start of treatment (Day 1 of Cycle 1) up to Month 15
  Disease-free survival is the time until the date of documentation of first progressive disease (PD) or death.
Overall Survival | Start of treatment (Day 1 of Cycle 1) up to Month 15
  Overall survival is defined as the time from the start of treatment until death (whatever the cause). Participants still alive will be censored at the moment of last visit or contact.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag G.m.b.H, Germany Clinical Trial, Study Director — Janssen-Cilag G.m.b.H
Locations (3):
- Germany (3):
  - Kiel
  - Regensburg
  - Stuttgart

REFERENCES:
- See also: Pilot study with bortezomib in combination with rituximab standard therapy in patients with relapsed or refractory follicular lymphoma and at least 2 previous therapies — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=1713&filename=CR010342_CSR.pdf